CLINICAL TRIAL: NCT02322684
Title: Bougie-guided Tracheal Tube Placement Through the Air-Q® Intubating Laryngeal Airway: Clinical Evaluation
Brief Title: Endotracheal Intubation Using a Bougie Through the Air-Q Intubating Laryngeal Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Yasser Mostafa Samhan, Professor, Theodor Bilharz Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TBRI-airq
Record Dates: First submitted 2014-12-15; First posted 2014-12-23 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Airway Complication of Anaesthesia
Keywords: Bougie; Air-Q; Insertion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Q (Active Comparator): Blind endotracheal intubation will be performed through the air-Q
  Interventions: Device: Air-Q
- Group B (Active Comparator): Blind endotracheal intubation will be performed through the air-Q with bougie assisted
  Interventions: Device: Air-Q

INTERVENTIONS:
Device: Air-Q — Air-Q/Intubating Laryngeal Airway (air-Q/ILA, Cookgas LLC, St. Louis, MO, USA) is an extra glottis airway (EGA) used as a primary airway device or as an adjunct to tracheal intubation. The air-Q/ILA is available as a disposable (air-Q) or nondisposable (ILA) device
  Other Names: Intubating laryngeal Airway

SUMMARY:
The purpose of this study is to assess the success rate of bougie-guided endotracheal intubation compared to blind intubation through the Air-Q intubating laryngeal mask

DETAILED DESCRIPTION:
After ethical committee approval and written informed consent, 140 patients of either sex, > 18 years old, ASA physical status I and II scheduled to receive general anesthesia with tracheal intubation for an elective surgical procedure will be enrolled in the study. They will be randomly allocated to one of two groups according to a computer generated list of 70 patients each. Blind endotracheal intubation will be performed through the air-Q with bougie assisted (Group B) or without assistance (Group Q). Patients ASA physical status >III, mouth opening <2 cm, increased risk of aspiration, those with poor lung compliance, with lesions of the oropharynx or epiglottis and known or anticipated difficult tracheal intubation or facemask ventilation will be excluded from the study.

In the operating room, the following monitors will be attached to the patients: five leads ECG, noninvasive blood pressure, pulse oximetry, ETCO2, anesthetic gas analyzer and neuromuscular monitoring (Infinity Kappa, Dräger, Lübeck, Germany). After adequate oxygenation, general anesthesia will be induced with 2 mg kg-1 propofol, 1-2 µg kg-1 fentanyl and 0.6 mg kg-1 rocuronium. Mask-ventilation with a mixture of oxygen and sevoflurane for an end-tidal concentration of 2% will be followed. The air-Q/ILA will be inserted once ulnar nerve train-of-four stimulation produced no visually detectable response while the patient's head in a neutral position. All airway manipulations (device insertion and tracheal intubation) will be performed by a senior anesthesiology staff member. The size of the air-Q will be selected on the basis of the patient's weight, in accordance with the corresponding manufacturer's recommendations. If ventilation with the device is unsatisfactory, the "Klein maneuver" corrects downfolding of the epiglottis by using a jaw thrust and an up-down maneuver of the ILA. During tracheal intubation through the air-Q/ILA, the tracheal tube is advanced to a depth of 12 to 15 cm so that the tip of the tube is close to the air-Q/ILA opening. Intubation through these supraglottic devices will be facilitated using a water-based lubricant. Then removal of the ILA immediately after tracheal intubation can be assisted by a stylet produced by the manufacturer. Tracheal intubation will be successful if ventilation through the tracheal tube produced an adequate chest expansion and a capnographic curve is obtained.

In group B, the operator gently inserts the bougie through the air-Q/ILA while looking at any bulges in the neck to judge the approximate positioning of the bougie. As soon as the bougie enters the trachea, a characteristic click is felt by the assistant and the operator feels the bougie entering in a hallow space. Another sign for intra tracheal bougie insertion when the bougie reaches the small bronchus between 30 and 40 cm marks (distal hold up sign). The air-Q/ILA is then removed and a tracheal tube is railroaded over the bougie.

Conventional single-use polyvinyl chloride (PVC) tracheal tubes (Mallinckrodt Company, Juarez, Chihuahua, Mexico) will be used for blind tracheal intubation in both groups: size 7.0 mm ID tracheal tubes for patients weighing ≥50 kg and 6.0 mm ID tubes for patients <50 kg. In both study groups, 3 attempts at device insertion and intubation will be allowed. Intubation will be only attempted if appropriate ventilation is obtained. Lung ventilation through the supraglottic device is permitted between intubation attempts. If tracheal intubation through the device is unsuccessful, it is performed by direct laryngoscopy.

The following parameters will be measured:

* Mallampati score, mouth opening (cm), thyromental distance (cm), neck circumference (cm)
* Air-Q™ /ILA insertion: insertion time (seconds), ease of insertion (easy, difficult), number of attempts, 1st attempt success rate and grade of ventilation (adequate, possible or impossible).
* Tracheal intubation: number of attempts, intubation time (seconds), 1st attempt success rate and overall success rate, ,
* Air-Q insertion time: is the time from introducing the device in mouth till attachment to the circuit and capnographic trace is obtained.
* Bougie insertion time: is the time from removal of the breathing circuit from air-Q to the feeling of hold up sign.
* ETT insertion time: is the time from insertion of the tracheal tube in the device until confirmation by capnographic trace.
* Total intubation time in group Q (air-Q™ /ILA insertion time plus intubation time) and the total intubation time in group B (air-Q™ /ILA insertion time plus bougie insertion time plus bougie guided intubation time) were calculated.
* We also recorded the types of and number of adjusting maneuvers for each attempt, frequency of esophageal intubation, and any incidence of hypoxia (SpO2<95%).
* Incidence of airway complications at insertion of air-Q™ /ILA, gum elastic bougie and ETT as trauma to mouth, lips or tongue and visible or occult blood.
* Incidence of Airway Morbidity at 18-24 h postoperatively in both groups as sore throat, dysphagia, dysphonia and its degree (mild/moderate/severe)
* Hemodynamic data heart rate (HR) and mean arterial blood pressure (MAP) were also recorded at the following time intervals:

T0, baseline before induction T1, before air-Q™ insertion T2, after air-Q™ insertion T3, before bougie insertion T4, after bougie insertion T5, before ETT insertion through the device T6, after ETT intubation T7, 1 min after intubation T8, 5 min after intubation T9, 10 min after intubation

Statistical Analysis

As no previous study researching bougie guided endotracheal intubation through air-Q™, we consider this research as a pilot study and 70 patients in each group is suitable. Results are expressed as mean ± standard deviation (SD) or number (%). Categorical data was compared using Chi square test. Variables in both groups were compared using either unpaired t test or Mann Whitney test whenever it was appropriate. Intra-group comparison (within group comparison) between mean values of variables measured at baseline and different times was performed using repeated measures ANOVA followed by Bonferroni test if significant results was recorded. Data analysis was performed using Statistical Package for Social Sciences (SPSS) version 19 computer program. Significance was considered when P-value ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* 19-60 years old,
* ASA physical status I and II
* Patients scheduled to receive general anesthesia with tracheal intubation for an elective surgical procedure.

Exclusion Criteria:

* Age <19 & >60
* ASA physical status ≥ III,
* Mouth opening <2 cm,
* Patients with increased risk of aspiration,
* Those with poor lung compliance,
* Patients with lesions of the oropharynx or epiglottis
* Patients known or anticipated to have difficult tracheal intubation or facemask ventilation.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Assess bougie-guided tracheal tube placement through the air-Q® Intubating Laryngeal Airway regarding success rate on the first attempt | Three attempts are allowed (up to 5 minutes)
  The operator gently inserts the bougie through the air-Q/ILA while looking at any bulges in the neck to judge the approximate positioning of the bougie. As soon as the bougie enters the trachea, a characteristic click is felt by the assistant and the operator feels the bougie entering in a hallow space. Another sign for intra tracheal bougie insertion when the bougie reaches the small bronchus between 30 and 40 cm marks (distal hold up sign). The air-Q/ILA is then removed and a tracheal tube is railroaded over the bougie.

SECONDARY OUTCOMES:
The overall success rate | 5 minutes
  The air-Q/ILA insertion and endotracheal insertion success rate (1st+2nd+3rd attempts)
The tracheal intubation time | 1 minute
  It is the calculated from the insertion of the tracheal tube in the device until confirmation of adequate lung ventilation

OTHER OUTCOMES:
The number of attempts | 5 minutes
  up to three attempts
Complications (Sore throat, dysphagia, dysphonia and its degree (mild/moderate/severe) | 24 hours
  Sore throat, dysphagia, dysphonia and its degree (mild/moderate/severe)

CONTACTS AND LOCATIONS:
Overall Officials: Reeham S. Ebied, M.D., Principal Investigator — Theodor Bilharz Research Institute
Locations (1):
- Theodor Bilharz Research Institute, Giza, Egypt

REFERENCES:
- See also: Theodor Bilharz Research Institute — http://www.tbri.sci.eg/